CLINICAL TRIAL: NCT00317265
Title: Complete Arterial Revascularization and Conventional Coronary Artery Surgery Study (CARACCASS)-European Multicenter Study
Brief Title: Coronary Bypass Surgery Trial: Complete Arterial Revascularization and Conventional Coronary Artery Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK NR-348/98
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coronary bypass surgery; complete arterial coronary surgery; internal mammary artery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

INTERVENTIONS:
Procedure: Coronary bypass surgery

SUMMARY:
This is a randomized, prospective European Multicenter Study comparing complete arterial revascularization of the coronary arteries using arterial graft material exclusively and "conventional" coronary artery bypass surgery using the left internal thoracic artery as graft to the left anterior descending artery (LAD) and vein grafts to other vessels to be bypassed.

DETAILED DESCRIPTION:
Coronary artery surgery effectively relieves angina and prolongs life in certain patient subsets. It is the most frequently performed major surgical procedure and therefore has profound economical impact. Unfortunately angina returns in 10 to 20 percent of patients by five years and in up to 50 percent at 10 years primarily because of graft failure and progression of atherosclerosis in the native coronary arteries. Serial angiography reveals that 15-30 percent of vein grafts are stenosed at one year and that nearly 50 percent are occluded at ten years. Recurrence of angina is associated with an increased risk of late myocardial infarction and reoperation. Reoperations after cardiac surgery carry a significantly increased risk of morbidity and mortality due to increased patient age, progression of coronary atherosclerosis, frequently reduced left ventricular function and technical difficulties. Thus prevention of restenosis by medical and surgical means is of eminent importance.The use of the IMA as a graft to the LAD is proven to reduce long-term mortality in patients after CABG throughout a 15 year follow-up period in all age groups. This data and the further improved survival with bilateral IMA grafting suggested by some have increased the interest of the surgical community in total arterial revascularization using both IMAs and various other arterial conduits.

However to date there is no conclusive data demonstrating a clinical benefit of total arterial revascularization.Reports available on complete arterial revascularisation are either single institution / single surgeon, retrospective or non - randomized. Data on which we base our daily decision making is by and large from a different surgical period with different techniques used. Improved understanding of the pathogenic processes leading to graft occlusion have led to more rigorous use of antiplatelet drugs and lipid lowering which may significantly improve vein graft patency rates and slow or halt progression of native coronary artery atherosclerosis in the future.

The scientific hypotheses underlying this randomized multicenter trial are:

1. With respect to the primary outcome variable "total mortality" complete arterial revascularisation does not cause a significantly higher mortality over 5 years of follow-up (as compared to conventional coronary artery surgery) i.e. non-inferiority due to increased tecnical complexity of the surgical procedure.
2. In terms of the combined secondary outcome variable "cardiac death, nonfatal myocardial infarction and re-revascularisation (PTCA or CABG)" and additional outcome variables "freedom from angina, functional status and quality of life" complete arterial revascularisation shows a clear benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible for surgical myocardial revascularization
2. Age 70 years or less
3. Triple vessel coronary disease with significant coronary artery stenosis defined as a stenosis of at least 50% in luminal diameter
4. Patients with stable angina pectoris (Canadian Cardiovascular Society 1, 2, 3, or 4) or unstable angina pectoris (Braunwald Classification 1b, 2b, 3b) or proven silent myocardial ischemia.

Exclusion Criteria:

1. No informed consent
2. Age > 65 years
3. Participation in another study with any investigational drug or coronary revascularization procedure
4. When follow up over a period of five years is difficult or unlikely
5. Concomitant non-cardiac disease likely to limit long-term prognosis (e.g. cancer)
6. One or two vessel coronary disease and isolated left main stenosis
7. Estimated left ventricular ejection fraction < 25%
8. Myocardial infarction within seven days
9. Need for concomitant major cardiac or non-cardiac surgery (e.g. valve surgery, left ventricular aneurysm, aortic aneurysm, carotid artery desobliteration, etc.)
10. Redo-cardiac surgery
11. Presence of the combination of insulin dependent diabetes mellitus and chronic obstructive pulmonary disease requiring therapy
12. Renal insufficiency requiring dialysis
13. Presence of the combination of severe adiposity and insulin dependent diabetes mellitus
14. Presence of the combination of severe adiposity and chronic obstructive pulmonary disease requiring therapy
15. Severe hepatic disease
16. Emergent operation for coronary artery disease with signs of ischemia (e.g. failed PTCA, ongoing myocardial infarction)
17. Unstable angina pectoris Class A and C according to Braunwald classification (i.e. secondary unstable angina and postinfarction unstable angina within one week after acute MI)
18. Inadequate quality of saphenous vein material
19. Inadequate quality or number of arterial conduits to achieve complete revascularization likely (e.g. chest irradiation, major abdominal surgery)
20. Recent (< 2weeks) cerebrovascular event (TIA, RIND, stroke)

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 1999-01; Study Completion 2005-01

PRIMARY OUTCOMES:
All cause mortality perioperatively, one year, five and ten years.

SECONDARY OUTCOMES:
Combined cardiac death, non-fatal myocardial infarction and repeat revascularisation at one, five and ten years.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Simon, MD, Principal Investigator — Dept. of Cardiothoracic Surgery, Medical Univ. of Vienna
Locations (14):
- Austria (2):
  - Dept. of Surgery I, AKH Linz, Linz
  - Dept Cardiothoracic Surgery, Medical Univ. of Vienna, Vienna
- Czechia (2):
  - Clinic for Cardiovascular Surgery, IKEM, Prague
  - Kardiochirurgie, Nemocnice Podlesi, Třinec
- Germany (4):
  - Kerckhoff-Klinik, Bad Nauheim
  - Dept.of Cardiac Surg, Ruhr University, Bochum
  - Dept of Cardiothoracic and Vascular Surgery, J-W-Goethe University, Frankfurt
  - HKZ Rotenburg, Rothenburg An Der Fulda
- Hjerteklinikken St. Elisabeth, Regionsykehuset Trondheim, Trondheim, Norway
- Dept Cardiothoracic Surg, Univ. of Gdansk, Gdansk, Poland
- Spain (3):
  - Dept of Cardiovasc Surg, Hospital Clinico, University of Barcelona, Barcelona
  - Dept of Cardiac Surg, Hospital de Cruces, Bilbao
  - Dept. of Cardiovascular Surgery, University of Salamanca, Salamanca
- Department of Cardiothoracic Surgery, University Hospital, Linköping, Sweden